CLINICAL TRIAL: NCT03945552
Title: Universal Strengths-Based Parenting Support in Pediatric Health Care for Families With Very Young Children Following the Flint Water Crisis
Brief Title: Pediatric Parenting Support in Flint
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Michigan State University (Other); University of Michigan (Other); Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-01347; R01HD096909-01A1 (NIH)
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Family Research
Keywords: Parenting Practices; Parent-Child Relationships; Child Development

STUDY DESIGN:
Intervention Model Description: Approximately 600 potential infant/parent dyads screened for inclusion and exclusion criteria.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Care as usual
- Video Interaction Project (Experimental): VIP is a strengths-based, family-centered intervention that uses pediatric well-child visits to enhance parenting practices/relationships and child development by promoting positive parenting practices such as pretend play, shared reading, and daily routines.
  Interventions: Behavioral: Video Interaction Project

INTERVENTIONS:
Behavioral: Video Interaction Project — VIP is a strengths-based, family-centered intervention that uses pediatric well-child visits to enhance parenting practices/relationships and child development by promoting positive parenting practices such as pretend play, shared reading, and daily routines.
  Arms: Video Interaction Project

SUMMARY:
Public health disasters have disproportionate impacts on low income communities, through pathways that add to those of poverty and associated stressors, and act over extended periods. Very young children are highly vulnerable to long-term impacts on development and mental health in the context of parenting challenges following disasters, yet frequently receive the least attention and resources. This study will test the role of universal parenting support in enhancing young children's development and mental health in Flint, Michigan following the Flint Water Crisis.

DETAILED DESCRIPTION:
There are three specific aims of this study: Specific Aim 1: Characterize participants' experience of the FWC using ecological (neighborhood-level), geocoded STYH data, ecological indicators of water quality and parent self-report measures. These metrics will be obtained from Speak to Your Health (STYH) survey, a biennial community survey including neighborhood-level measures of stress collected before, during and after the FWC. Specific Aim 2: Assess impacts of strengths-based parenting support (VIP) after a disaster compounding chronic poverty (FWC). Specific Aim 3: Assess variation in VIP impacts in relation to FWC experience.

ELIGIBILITY:
Inclusion Criteria:

* Infant is receiving pediatric care at Hurley Children's Clinic
* Caregiver can be contacted (has a working phone)
* Infant is three months old or younger at time of enrollment

Exclusion Criteria:

* Infant very low birth weight (<1500gm)
* Infant born in non-singleton birth (twin, triplet, etc.)
* Infant has known or suspected significant genetic syndrome or malformation
* Infant has other significant medical or developmental complication or risk (e.g., known neurodevelopmental/neuromuscular disorder likely to affect development)
* Parent/legal guardian not present with infant at visit and/or unable to provide consent
* Parent/legal guardian is not English speaking
* Parent/legal guardian with known significant impairment that will be barrier to communication and participation (e.g., intellectual disability, schizophrenia)
* Parent/legal guardian has previously participated in VIP intervention with another child
* Not planning to stay in Flint area for at least 3 years

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
Parenting compensatory factors (Assets/vulnerabilities): Parenting Stress | 6 months to 4 years
  Parenting stress measured by Parent Survey (PS) with the Parenting Stress Index (PSI; α= .82) short form parental distress subscale, range 12-60, higher scores worse.
Positive Parenting Activities | 6 months to 4 Years
  Positive parenting practices measured by parent survey (PS) with the StimQ2's core subscales: Reading (READ), Teaching (Parental Involvement in Developmental Advance), and Responsivity (Parental Verbal Responsivity) Subscales. The StimQ2 is a structured interview. The three subscales are summed to obtain a total score. Total scores can range from 0 to 42 (infant)/46 (toddler)/60 (preschool). Higher score better.
Parent-child Interaction and relationship | 6 months to 4 Years
  Laboratory observation of semi-structured interactions with real time Parenting Interactions with Children: Checklist of Observations Linked to Outcome (PICCOLO), and Adult-Child Interactive Reading Inventory (ACIRI) coding.
Child Expressive and Receptive Language Development | 6 months to 4 Years
  Measured through direct assessment of child using the Mullen Scales of Early Learning. The Mullen provides standardized scores (M=50, SD=10). Higher scores better.
Child Social-Emotional Development | 18 months to 4 years
  Measured by parent survey (PS) using the Infant-Toddler Social Emotional Assessment (ITSEA). ITSEA is a structured interview that measures 4 domains. Items have a 3-point response scale. Subscales are scored by taking the average of items, and subscales are then added to create an overall score. Scores are standardized on a T-distribution (M=50, SD=10). Higher scores worse, except for Competence domain.

SECONDARY OUTCOMES:
Parent Self-Efficacy Measured by the Parent Reading Beliefs Inventory (PRBI) | birth to 4 years
  Self-efficacy measured by parent survey (PS) using the Parent Reading Beliefs Inventory (PRBI), Teaching Efficacy subscale (α=.73). PRBI is a structured interview. Items are rated on a 1 to 4 Likert scale. Scores for Teaching Efficacy range from 9 to 36. Higher scores are better.
Parent Self-Efficacy Measured by the Parenting Self Agency Measure (PSAM) | birth to 4 years
  Parenting self-agency measured by PS using the Parenting Self-Agency Measure (PSAM). PSAM is a 5-item questionnaire, with items rated from 1 to 5. Scores range from 5 to 25. Higher scores are better
Parent Self-Efficacy Measured by Resiliency (RSA) | birth to 4 years
  Resiliency measured using the Resiliency Scale for Adults (RSA), Personal Strength and Social Resources subscales. RSA items are scored on a 1 to 5 Likert scale. Subscale scores are averaged across items. Higher scores are better.
Parenting compensatory factors: Planning and Organization | 6 months to 4 years
  Feeding, sleeping, media routines and screen time measured by parent survey (PS) using an internal survey (PI Mendelsohn; kappa 0.91).
Parenting compensatory factors: Parenting Interaction Skills and Resources | 6 months to 4 years
  Play coded video for VIP-promoted skills measured using VIP observation checklist
Parent-child interactions and relationship | 6 months to 4 years
  Laboratory observation of semi-structured interactions with subsequent global coding using the Caregiver-Child Affect, Responsivity, and Engagement Scale (C-CARES) and the Parent Child early Relational Assessment (PCERA)
Naturalistic assessment of parent-child interaction | 6 months to 4 years
  LENA Home (adult words, conversational turns)
Negative Parenting Practices | 6 months to 4 years
  Socolar Discipline Survey (α= .56-.82) will be used to assess harsh discipline punishment. Answers range from 1 (never) to 6 (always), where a higher score indicates great frequency of harsh discipline. A total score is calculated from the sum of all items.
Child naturalistic language/narrative development | 18 months to 4 years
  Laboratory observation of naturalistic assessment of child language/narrative
Child self-regulation | 18 months to 4 years
  Direct observation using subset of executive function (EF) battery for 3-year olds from S.M. Carlson - Dimensional Card Sort (3 incompatible test trials, scored 0/1), Fruit Stroop (mismatched fruit; 3 trials, scored 0-2), and Bear/Dragon: Go/No Go (10 trials, scored 0/1).
  Laboratory observation of child regulation during assessment using the Preschool Self-Regulation Assessment (PSRA).

CONTACTS AND LOCATIONS:
Overall Officials: Alan Mendelsohn, MD, Principal Investigator — New York Langone Medical Center
Locations (2):
- United States (2):
  - Hurley Children's Hospital, Flint, Michigan
  - New York University School of Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Given that the proposed research methodology will take place in a community (Flint, MI) with ongoing institutional mistrust following the onset of a community-level disaster (the Flint Water Crisis), the investigators are committed to developing a plan for data sharing that will meet NIH's data sharing requirements while simultaneously meeting the needs of this community. The investigators will work together with the Michigan State University Pediatric Public Health Initiative and its community partners to develop a plan for data sharing that addresses these diverse and important considerations.
Supporting Information: Study Protocol
Time Frame: Data will become available after all primary outcomes have been assessed by study investigators. Time frame for availability of data will depend of other researchers' specific requests and community partners needs.
Access Criteria: Researchers from accredited academic institutions may request access to the study protocol. Permission and access will be granted on an ad hoc basis.

REFERENCES:
- [Derived] Chen Y, Canfield CF, Finegood ED, Gutierrez J, Williams S, O'Connell LK, Mendelsohn A. Family stress model and parenting in infancy: Social support and parenting self-efficacy as resilience factors. J Fam Psychol. 2025 Dec;39(8):1129-1140. doi: 10.1037/fam0001341. Epub 2025 Aug 14. PMID 40811117